CLINICAL TRIAL: NCT02268149
Title: The Effect of Multiple Doses of BIIL 284 BS on the Pharmacokinetics of a Single Dose of Prednisone in Healthy Male Subjects (A Randomized, Double-blind, Placebo-controlled, Two Period, Two-way Cross-over Study)
Brief Title: Study to Evaluate the Effect of Multiple Doses of BIIL 284 BS on the Pharmacokinetics of Prednisone in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 543.24
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — amelubant; Prednisone

ARMS (2):
- BIIL 284 BS + Prednisone (Experimental): BIIL 284 BS 9 days; prednisone 2 single doses
  Interventions: Drug: BIIL 284 BS; Drug: Prednisone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIL 284 BS
  Arms: BIIL 284 BS + Prednisone
Drug: Prednisone
  Arms: BIIL 284 BS + Prednisone
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to evaluate the effect of multiple doses of BIIL 284 BS on the pharmacokinetics of a single dose of prednisone

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed and dated prior to participation into the study
* All participants in the study should be healthy males, aged 18-50 years old inclusive
* All participants should be within (+- 20%) of their ideal body weight (Broca-Index)
* Non-smokers (subject who have never smoked) or ex-smoker for at least one year with a smoking history, no greater than five pack-years (1 pack year = 20 cigarettes per day for 1 year)
* Ability to comply with the concomitant therapy restrictions as detailed in Clinical Trial Protocol (CTP)
* Subjects will be off all prescription drugs. O.T.C. drugs must be discontinued for at least two weeks prior to participation in the study. If throughout the study, subjects need any O.T.C. medication, the investigator will call the clinical monitor and this will be reviewed on a case-by-case basis. Restrictions for different medications are described in CTP
* Subjects will have no evidence of clinically relevant concomitant disease based upon complete medical history, full physical examination, chest-x-ray (if not done in previous 6 months), ECG and clinical laboratory tests

Exclusion Criteria:

* Viral respiratory tract infection or a respiratory tract infection within the six weeks preceding dosing with study medication
* Small or difficult to locate arm or hand veins that would impair the clinicians ability to draw blood samples or to place a venous catheter
* Subjects with a known drug or alcohol dependence (absence of dependency for 10 years) or who drink more than 60 g of alcohol per day, history of significant allergic reactions to drugs or sensitivity to aspirin or positive drug screen
* Use of investigational new drug in the preceding month or six half-lives (whichever is greater) prior to the first screen at Visit 1
* Donation of blood during the month preceding Visit 1
* Subjects receiving hyposensitization therapy who are not on a stable dose for the last three months before Visit 1
* Subjects with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Subjects with diseases of the central nervous system (such as epilepsy) or with psychiatric disorders
* Subjects with known history of orthostatic hypotension, fainting spells or blackouts
* Subjects with chronic or relevant acute infections
* Subjects with history of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Subjects with eosinophilia > 7 %
* Subjects who received any other drugs, which might influence the results of the trial during the weeks prior to dosing with study medication
* Subjects who participated in excessive physical activities (e.g. competitive sports) within the last week before dosing with study medication

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2000-04; Primary Completion 2000-07 (Actual)

PRIMARY OUTCOMES:
AUC (Area under the concentration-time curve of the analyte in plasma) | up to 72 hours post dose
Cmax (Maximum measured concentration of the analyte in plasma) | up to 72 hours post dose
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 72 hours post dose
t½ (Terminal half-life of the analyte in plasma) | up to 72 hours post dose
MRTtot (total Mean residence time) | up to 72 hours post dose
CLtot/F (Total clearance of the analyte in plasma after oral administration) | up to 72 hours post dose
Vz/F (Apparent volume of distribution of the analyte during the terminal phase) | up to 72 hours post dose

SECONDARY OUTCOMES:
Number of subjects with adverse events | up to 53 days
Changes in immunomodulatory assessed by T-cell proliferation | predose, 4 hours post dose
Changes in Interleukin-2 (IL-2) levels | predose, 4 hours post dose
Changes in Interferon gamma (IFNy) levels | predose, 4 hours post dose